CLINICAL TRIAL: NCT00283309
Title: Memantine or Riluzole Prophylaxis for Corticosteroid-induced Mood and Declarative Memory Changes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study finished enrollment but data was never sent for publishing.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Principal Investigator, MD/PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 042005-018
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Mood; Memory Deficit
Keywords: Corticosteroids; Riluzole; Memantine; Memory
MeSH Terms: conditions — Memory Disorders | interventions — Memantine; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Memantine (Active Comparator): Memantine is used to determine if patients given pretreatment to corticosteroid therapy for inflammatory illnesses will show lesser declarative memory impairment than those receiving placebo. Baseline 10mg x 3 days, then 10mg BID x 4 days.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Inactive ingredient matching the active medication in appearance
  Interventions: Drug: Memantine; Drug: Riluzole
- Riluzole (Active Comparator): Riluzole is given to patients receiving corticosteroid therapy for inflammatory illnesses pretreatment to determine if they show lesser declarative memory impairment than those receiving placebo. Baseline 50mg x 3 days, then 50mg BID x 4 days.
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Memantine
  Arms: Memantine; Placebo
Drug: Riluzole
  Arms: Placebo; Riluzole

SUMMARY:
The primary purpose is to determine if patients scheduled to receive prescription corticosteroid therapy for inflammatory illnesses who are given either memantine or riluzole pretreatment will show lesser declarative memory impairment than those receiving placebo.

The exploratory purpose is to determine if patients scheduled to receive prescription corticosteroid therapy for inflammatory illnesses who are given memantine or riluzole pretreatment will show a smaller increase in manic/hypomanic symptom severity than those receiving placebo.

DETAILED DESCRIPTION:
Twenty five (25) outpatients with pulmonary (e.g. asthma, cystic fibrosis) or rheumatic (e.g. rheumatoid arthritis, dermatomyositis) illnesses scheduled to receive a brief course ("burst") of prednisone will be enrolled. The subjects will be randomized to receive memantine, riluzole or placebo beginning immediately prior to the corticosteroid therapy and continuing for one week. Measures of cognition and mood will be compared between the two groups at baseline, day 3, and day 7.

Demographic information including age, gender, frequency and duration of prior corticosteroid therapy and current anticipated dose and duration will be collected at baseline. Baseline measures of mood will be assessed with the Activation subscale of the Internal State Scale (ISS) (primary measure), Hamilton Depression Rating Scale (17-item version), and Young Mania Rating Scale (YMRS). Cognition will be assessed with the RAVLT (primary measure), Stroop, and Digit Span Backwards. The subjects will be given memantine (10 mg), riluzole (50 mg), or identical appearing placebo 1 tablet daily for 3 days and then at the first follow up appointment (day 3) the dose will be increased to BID if no side effects are reported. The subjects will be reassessed twice, at day 3 and day 7. Mood and cognitive measures will be repeated. The study visits will last approximately an hour and a half. Participants will discontinue memantine when they discontinue prednisone. The RA administering assessments will be blinded at all times. Alternative but equivalent versions of the RAVLT and Digit Span Backwards will be given to minimize practice or learning effects. Current and cumulative corticosteroid dose (mg each day X number of days) will be determined and recorded.

HVLT-R test total words recalled scores will be compared between baseline and exit of the active medication phase and placebo phase using a within subjects design and paired t-tests. Based on our prior experience working with corticosteroid-dependent patients we have found them to be very compliant with clinical treatment. Thus, we do not anticipate large numbers of dropouts or missing data. In the case of missing data we will use the last observation carried forward. In our lamotrigine study in a similar population, we found a change in total words recalled on a word list and on the Stroop. Assuming a similar change with memantine, using double-sided, paired t-tests, we could detect a difference with a change in the placebo group with participants on the HVLT-R and up to with participants on the Stroop. Thus, although this is primarily a pilot study to obtain effect sizes for future, larger trials funded by NIH, it should have power to detect clinically meaningful differences between medication and placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* English speaking
* Able to provide informed consent
* Scheduled to receive a corticosteroid burst of at least 20 mg prednisone or equivalent for at least 7 days

Exclusion Criteria:

* History of allergic reaction to memantine and/or riluzole
* Pregnant or nursing women
* History of liver disease, myocardial infarction, renal failure, diabetes with poor glycemic control, or other unstable medical condition
* Mental retardation, dementia, or other severe cognitive disorder
* Prior prednisone therapy in the last 14 days
* Current alcohol/substance abuse/dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern, Dallas, Texas, United States